CLINICAL TRIAL: NCT01487161
Title: A Double-Blind, Randomized, Parallel Group, Dose-Ranging Study Comparing FX006 to Commercially Available Triamcinolone Acetonide Injectable Suspension in Patients With Osteoarthritis of the Knee
Brief Title: Study of FX006 in Patients With Osteoarthritis of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FX006-2011-001
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: osteoarthritis; knee; pain; corticosteroid; intra-articular; injection
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — FX006; Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FX006 10 mg (Experimental): Single 3 mL intra-articular (IA) injection Extended-Release Formulation
  Interventions: Drug: FX006
- FX006 40 mg (Experimental): Single 3 mL intra-articular (IA) injection Extended-Release Formulation
  Interventions: Drug: FX006
- FX006 60 mg (Experimental): Single 3mL intra-articular (IA) injection Extended-Release Formulation
  Interventions: Drug: FX006
- TCA IR 40 mg (Active Comparator): Single 1 mL intra-articular (IA) injection Immediate-Release Triamcinolone Acetonide
  Interventions: Drug: TCA IR

INTERVENTIONS:
Drug: FX006 — Single 3 mL intra-articular injection
  Arms: FX006 10 mg; FX006 40 mg; FX006 60 mg
Drug: TCA IR — Single 1 mL intra-articular injection
  Other Names: Kenalog®-40 Injection; Kenacort-A 40; Triamcinolone Acetonide Crystalline Suspension (TAcs)
  Arms: TCA IR 40 mg

SUMMARY:
The purpose of this study was to evaluate the safety, efficacy and pharmacokinetics of FX006 in patients with osteoarthritis of the knee.

DETAILED DESCRIPTION:
Study FX006-2011-001 was a multi-center, randomized, double-blind, active comparator, parallel-group, single-dose study designed to assess the magnitude and duration of pain relief of three doses (10, 40, and 60 mg) of FX006, an extended-release formulation of TCA, relative to commercially-available TCA IR.

The general tolerability of a single injection of FX006 also was assessed.

Secondary objectives included exploration of the effect of FX006 on functional improvement, responder status, time to onset of pain relief, global impressions of change, and consumption of analgesic medications and evaluation of the PK profile of single injection of the three dose levels of FX006.

The study was planned to be conducted in up to 224 male and female patients ≥40 years of age with OA of the knee enrolled at 22 study centers in the US, Australia, and Canada.

ELIGIBILITY:
Main Inclusion Criteria:

* Willingness and ability to comply with the study procedures and visit schedules and ability to follow verbal and written instructions
* Male or female >=40 years of age
* Diagnosis of unilateral or bilateral OA of the knee for at least 6 months prior to Screening with confirmation of OA according to American College of Rheumatology Criteria for Classification of Idiopathic OA of the Knee (clinical and radiological) based on an X-ray performed within 6 months prior to Screening or during the Screening period
* Qualifying mean score on the 24-h average pain score (0-10 numeric rating scale)
* Body mass index (BMI) ≤ 40 kg/m2
* Willingness to abstain from use of restricted medications

Main Exclusion Criteria

* Ipsilateral hip OA
* Fibromyalgia, chronic pain syndrome or other concurrent medical or arthritic conditions which could interfere with the evaluation of the index knee
* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, arthritis associated with inflammatory bowel disease, sarcoidosis or amyloidosis
* History of arthritides due to crystals (e.g., gout, pseudogout)
* History of infection in the index joint
* Clinical signs and symptoms of active knee infection or crystal disease of the index knee
* Presence of surgical hardware or other foreign body in the index knee
* Unstable joint (such as a torn anterior cruciate ligament)
* IA corticosteroid (investigational or marketed) in any joint within 3 months of Screening
* IA hyaluronic acid (investigational or marketed) in the index knee within 6 months of Screening
* Oral, inhaled and intranasal corticosteroids (investigational or marketed) within 1 month of Screening
* Prior arthroscopic or open surgery of the index knee within 12 months of Screening
* Planned/anticipated surgery of the index knee during the study period
* Active or history of malignancy within the last 5 years, with the exception of resected basal cell carcinoma, squamous cell carcinoma of the skin, or resected cervical atypia or carcinoma in situ
* Insulin-dependent diabetes
* Active psychiatric disorder including psychosis and major depressive disorder
* History of or active Cushing's syndrome
* Any other clinically significant acute or chronic medical conditions (e.g., uncontrolled diabetes)
* Skin breakdown at the knee where the injection would take place
* Women of child-bearing potential not using effective contraception or who are pregnant or nursing

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil Bodick, MD, PhD, Study Director — Flexion Therapeutics
Locations (21):
- United States (2):
  - Tucson, Arizona
  - Duncansville, Pennsylvania
- Australia (9):
  - Broadmeadow, New South Wales
  - Kogarah, New South Wales
  - St Leonards, New South Wales
  - Wollongong, New South Wales
  - Kippa-Ring, Queensland
  - Maroochydore, Queensland
  - Sherwood, Queensland
  - Clayton, Victoria
  - Malvern East, Victoria
- Canada (10):
  - Halifax, Nova Scotia
  - Etobicoke, Ontario
  - Newmarket, Ontario
  - Saint Catherine's, Ontario
  - Sarnia, Ontario
  - Thornhill, Ontario
  - Waterloo, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec

REFERENCES:
- See also: Journal of Bone & Joint Surgery - American Volume: 3 June 2015 - Volume 97 - Issue 11 - p 877-888 — http://journals.lww.com/jbjsjournal/Abstract/2015/06030/An_Intra_Articular,_Extended_Release_Formulation.1.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study took place at 22 centers across the United States, Canada and Australia. Enrollment took approximately 7 months.
Pre-assignment Details: Subjects were screened within 21 days of being randomized
Groups:
- FX006 10 mg: 58 subjects received FX006 10 mg as a single 3 mL IA injection.
- FX006 40 mg: 59 subjects received FX006 40 mg as a single 3 mL IA injection.
- FX006 60 mg: 60 subjects received FX006 60 mg as a single 3 mL IA injection.
- TCA IR (40 mg): 51 subjects received TCA IR 40 mg as a single 1 mL IA injection.
Period: Overall Study
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR (40 mg)
Started | 58 | 59 | 60 | 52
Completed | 56 | 57 | 59 | 50
Not Completed | 2 | 2 | 1 | 2
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 2
Not completed — missing data | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: A total of 229 patients were randomized to treatment in this study. 228 of 229 randomized patients received treatment and were included in the Safety Population; 1 patient randomized to the TCA IR group withdrew consent before receiving study treatment and was excluded.
Groups:
- FX006 10 mg; FX006 40 mg; FX006 60 mg: Single 3 mL IA injection
- TCA IR (40 mg): Single 1 mL IA injection
- Total: Total of all reporting groups
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR (40 mg) | Total
Number analyzed (Participants) | 58 | 59 | 60 | 51 | 228
Age, Continuous [Mean (Full Range); unit: years] | 61.5 [43 to 82] | 60.9 [40 to 80] | 61.9 [44 to 86] | 61.6 [42 to 83] | 61.5 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 31 | 34 | 29 | 120
  Male | 32 | 28 | 26 | 22 | 108

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Weekly Mean of the Average Daily (24-hour) Pain Intensity Score for FX006 60 mg vs TCA IR 40 mg
Description: The pain intensity score is measured using an 11-point numeric rating scale (NRS), where 0 indicates "no pain" and 10 indicates "pain as bad as you can imagine."
Time Frame: 8 weeks
Population: All patients who receive study treatment and have baseline and at least 1 post-dose pain evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- FX006 60 mg: FX006: Single 3 mL IA injection
- TCA IR 40 mg: TCA IR: Single 1 mL IA injection
Arm/Group | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 56 | 43
units on a scale | -3.9 (0.28) | -3.4 (0.31)
Statistical Analysis 1: Comparison: FX006 60 mg vs TCA IR 40 mg; Test type: Superiority; p = 0.1249, Longitudinal mixed effect model; Mean Difference (Final Values) = -0.5, 90% CI 2-sided [-1.2 to 0.2]

2. Primary Outcome: Change From Baseline to Week 10 in Weekly Mean of the Average Daily (24-hour) Pain Intensity Score for FX006 60 mg vs TCA IR 40 mg
Description: as for outcome 1
Time Frame: 10 weeks
Population: All patients who receive study treatment and have baseline and at least 1 post-dose pain evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 56 | 45
units on a scale | -3.6 (0.28) | -3.3 (0.31)
Statistical Analysis 1: Comparison: FX006 60 mg vs TCA IR 40 mg; Test type: Superiority; p = 0.2002, Longitudinal mixed effect model; Mean Difference (Final Values) = -0.4, 90% CI 2-sided [-1.1 to 0.3]

3. Primary Outcome: Change From Baseline to Week 12 in Weekly Mean of the Average Daily (24-hour) Pain Intensity Score for FX006 60 mg vs TCA IR 40 mg
Description: as for outcome 1
Time Frame: 12 weeks
Population: All patients who receive study treatment and have baseline and at least 1 post-dose pain evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 53 | 41
units on a scale | -3.2 (0.30) | -3.3 (0.33)
Statistical Analysis 1: Comparison: FX006 60 mg vs TCA IR 40 mg; Test type: Superiority; p = 0.5541, Longitudinal mixed effect model; Mean Difference (Final Values) = 0.1, 90% CI 2-sided [-0.7 to 0.8]

4. Secondary Outcome: Change From Baseline to Each of Weeks 8, 10, and 12 in Weekly Mean of the Average Daily (24-hour) Pain Intensity Score for FX006 10mg and 40 mg vs TCA IR 40 mg
Description: as for outcome 1
Time Frame: Weeks 8, 10 and 12
Population: All patients who receive study treatment and have baseline and at least 1 post-dose pain evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- FX006 10 mg; FX006 40 mg: FX006: Single 3 mL IA injection
Arm/Group | FX006 10 mg | FX006 40 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 51
units on a scale
  8 Weeks: number analyzed (Participants) | 55 | 55 | 43
  8 Weeks | -3.9 (0.28) | -4.3 (0.28) | -3.4 (0.31)
  10 Weeks: number analyzed (Participants) | 52 | 57 | 45
  10 Weeks | -3.8 (0.29) | -4.1 (0.29) | -3.3 (0.31)
  12 Weeks: number analyzed (Participants) | 48 | 43 | 41
  12 Weeks | -3.6 (0.30) | -3.7 (0.30) | -3.3 (0.33)

5. Secondary Outcome: Change From Baseline to Each of Weeks 1, 2, 3, 4, 5, 6, 7, 9, and 11 in Weekly Mean of the Average Daily (24-hour) Pain Intensity Score.
Description: as for outcome 1
Time Frame: Weeks 1-7 and Week 9 and 11
Population: All patients who receive study treatment and have baseline and at least 1 post-dose pain evaluation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 60 | 51
units on a scale
  Week 1: number analyzed (Participants) | 58 | 59 | 60 | 50
  Week 1 | -2.7 (0.24) | -3.0 (0.24) | -3.0 (0.24) | -3.1 (0.26)
  Week 2: number analyzed (Participants) | 57 | 59 | 60 | 49
  Week 2 | -3.6 (0.27) | -3.9 (0.27) | -3.8 (0.27) | -3.5 (0.29)
  Week 3: number analyzed (Participants) | 54 | 57 | 60 | 50
  Week 3 | -3.7 (0.27) | -4.1 (0.27) | -4.2 (0.27) | -3.5 (0.29)
  Week 4: number analyzed (Participants) | 56 | 56 | 60 | 47
  Week 4 | -3.8 (0.26) | -4.3 (0.26) | -4.2 (0.26) | -3.7 (0.28)
  Week 5: number analyzed (Participants) | 57 | 56 | 58 | 47
  Week 5 | -3.9 (0.28) | -4.3 (0.27) | -4.2 (0.27) | -3.5 (0.30)
  Week 6: number analyzed (Participants) | 58 | 56 | 56 | 49
  Week 6 | -4.0 (0.28) | -4.3 (0.28) | -4.2 (0.28) | -3.4 (0.30)
  Week 7: number analyzed (Participants) | 56 | 56 | 56 | 47
  Week 7 | -3.9 (0.28) | -4.4 (0.28) | -3.9 (0.27) | -3.3 (0.30)
  Week 9: number analyzed (Participants) | 53 | 54 | 57 | 45
  Week 9 | -3.8 (0.30) | -4.2 (0.30) | -3.7 (0.29) | -3.3 (0.32)
  Week 11: number analyzed (Participants) | 52 | 55 | 51 | 43
  Week 11 | -3.7 (0.30) | -3.9 (0.30) | -3.2 (0.29) | -3.4 (0.32)

6. Secondary Outcome: WOMAC A (Pain Subscale) Change From Baseline at Week 8
Description: The Western Ontario and McMaster Universities (WOMAC®) Osteoarthritis Index is a questionnaire that measures pain, stiffness, and function both independently and collectively, using a Likert 3.1, 5-point scale. The Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme, corresponding to an ordinal scale of 0-4. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 60 | 47
units on a scale | -1.23 (0.099) | -1.33 (0.098) | -1.16 (0.097) | -0.96 (0.108)

7. Secondary Outcome: WOMAC A1 (Pain on Walking Question) Change From Baseline at Week 8
Description: as for outcome 6
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- TCA IR 40 mg: FX006: Single 1 mL IA injection
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 60 | 47
units on a scale | -1.2 (0.12) | -1.2 (0.12) | -1.1 (0.11) | -0.8 (0.13)

8. Secondary Outcome: WOMAC B (Stiffness Subscale) Change From Baseline at Week 8
Description: as for outcome 6
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- TCA IR (40 mg): TCA IR: Single 1 mL IA injection
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR (40 mg)
Number analyzed (Participants) | 58 | 59 | 60 | 47
units on a scale | -1.37 (0.113) | -1.49 (0.112) | -1.24 (0.111) | -0.99 (0.124)

9. Secondary Outcome: WOMAC C (Function Subscale) Change From Baseline at Week 8
Description: as for outcome 6
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 58 | 60 | 47
units on a scale | -1.22 (0.096) | -1.31 (0.096) | -1.13 (0.095) | -0.94 (0.106)

10. Secondary Outcome: Percent of Responders According to OMERACT-OARSI Criteria at Week 8
Description: Outcome Measures in Rheumatoid Arthritis Clinical Trials - Osteoarthritis Research Society International. Responders are defined as participants with high improvement in pain or function.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 57 | 59 | 59 | 46
Participants | 52 | 53 | 47 | 32

11. Secondary Outcome: Responder Status as Defined by the Proportion of Patients Achieving >50% Improvement From Baseline in the Mean Daily Pain Intensity Scores at Week 8
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 55 | 55 | 56 | 43
Participants | 35 | 40 | 34 | 23

12. Secondary Outcome: Responder Status as Defined by the Proportion of Patients Achieving >30% Improvement From Baseline in the Mean Daily Pain Intensity Scores at Week 8
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 55 | 55 | 56 | 43
Participants | 42 | 47 | 45 | 27

13. Secondary Outcome: Responder Status as Defined by the Proportion of Patients Achieving >20% Improvement From Baseline in the Mean Daily Pain Intensity Scores at Week 8
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 55 | 55 | 56 | 43
Participants | 47 | 49 | 48 | 30

14. Secondary Outcome: Patient Global Impression of Change Scores at Week 8
Description: The Patient Global Impression of Change is a scale that aims to evaluate all aspects of participants' (patients') health and determining if there has been an improvement or not. The participant selects the one response from the response options that gives the most accurate description of his/her state of health (overall status). This is a 7-point scale, and scores range from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status.
Time Frame: Week 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 60 | 48
units on a scale | 1.9 (0.16) | 1.8 (0.16) | 2.4 (0.16) | 2.5 (0.17)

15. Secondary Outcome: Clinical Global Impression of Change Scores at Week 8
Description: The Clinical Global Impression of Change is a scale that the clinician uses to assess the participants' global function and determine if there has been an improvement or not. The clinician selects one response from the response options that gives the most accurate description of the participant's state of health (overall status). This is a 7-point scale, and scores range from 1 (Very Much Improved) to 7 (Very Much Worse). Lower scores indicate better health status.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 60 | 48
units on a scale | 1.9 (0.16) | 1.8 (0.16) | 2.5 (0.16) | 2.6 (0.17)

16. Secondary Outcome: Average Weekly and Total Consumption of Rescue Medications Over 8 Weeks.
Time Frame: 8 weeks
Measure: Least Squares Mean (Standard Error); unit: tablets (1tablet= 500 mg)
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR 40 mg
Number analyzed (Participants) | 58 | 59 | 60 | 48
tablets (1tablet= 500 mg) | 1.0 (0.22) | 1.0 (0.22) | 1.1 (0.22) | 1.2 (0.24)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from post injection on Day 1 through Day 85
Arm/Group | FX006 10 mg | FX006 40 mg | FX006 60 mg | TCA IR (40 mg)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59 | 0/60 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/58 | 2/59 | 1/60 | 0/51
Other Adverse Events (participants affected / at risk) | 13/58 | 16/59 | 22/60 | 22/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 10 mg (N=58) | FX006 40 mg (N=59) | FX006 60 mg (N=60) | TCA IR (40 mg) (N=51)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 10 mg (N=58) | FX006 40 mg (N=59) | FX006 60 mg (N=60) | TCA IR (40 mg) (N=51)
Nasopharyngits (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 7 (7) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Blood Glucose Increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Neutrophil Count Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
White Blood Cell Count Inreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Arthalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 8 (8) | 4 (4) | 2 (2)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 1 (1) | 5 (5) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes